CLINICAL TRIAL: NCT06811428
Title: Neonatal Comfort Seat Allowing Safe Lumbar Puncture and Minimizing Failure: a Randomized Controlled Trial
Acronym: NeoCALM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Joel Cox (Other)
Collaborators: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor-Investigator, Joel Cox, Dr. Joel Cox, MD, FRCPC, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LPCSRCT2025
Record Dates: First submitted 2025-01-31; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-01

CONDITIONS: Sepsis; Meningitis
Keywords: Lumbar puncture; Seating device; Positioning device; Newborn; Neonatal; Meningitis; Sepsis
MeSH Terms: conditions — Sepsis; Meningitis | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lumbar Puncture Comfort Seat Arm (Experimental): This is the group that will have the lumbar puncture conducted in an upright sitting position assisted by the medical device
  Interventions: Device: A novel device for immobilization of babies undergoing upright LP, the present working name (non-proprietary) for the device is LP Comfort Seat (LPCS)
- Standard of Care Arm (Active Comparator): This is the group that will have the lumbar puncture conducted in an upright sitting position assisted by the human assistant which is present standard of care
  Interventions: Other: Standard of Care (SOC)

INTERVENTIONS:
Device: A novel device for immobilization of babies undergoing upright LP, the present working name (non-proprietary) for the device is LP Comfort Seat (LPCS) — The participant will be placed in the LPCS for their lumbar puncture procedure
  Arms: Lumbar Puncture Comfort Seat Arm
Other: Standard of Care (SOC) — The patient will be held in the upright position by a human assistant
  Arms: Standard of Care Arm

SUMMARY:
A research trial which compares standard of care against employing a novel device for immobilization of babies undergoing upright LP, the present working name for the device is LP Comfort Seat (LPCS).

The research question is:

P: In late-preterm to term babies who are 0-28 days and undergoing LP for R/O Sepsis I: Is the LPCS more effective C: Than human/RN assisted upright positioning O: In generating a higher rate of first attempt LP success

Primary outcome measure is first attempt LP success (any evidence of CSF which is diagnostically useful by content and volume)

Secondary outcome measures could include

1. A qualitatively unadulterated tap (no blood) although as you know this is hard to control even with perfect positioning and technique and single pass
2. A difference in FLACC score as measure of overall pain/comfort between test and control

DETAILED DESCRIPTION:
Lay Description: Newborn babies who are unwell sometimes need to undergo a medical procedure known as a 'lumbar puncture' (also called 'spinal tap'). During this procedure, a needle is inserted at the base of the spine to extract fluid from the spinal column. This is most often done to determine if the baby has meningitis. The medical device presented here places the child's comfort and safety at the center of the spinal tap/ lumbar puncture experience and in doing increases the success of this otherwise stressful and technically challenging procedure. This is achieved by placing the child in a stable, firm, but comfortable position nearly eliminating patient motion which otherwise interferes with procedure success, and reduces the variability associated with a human assistant/holder

In the course of routine medical care of infants and young children, it may be necessary to conduct a procedure known as a 'lumbar puncture' or 'spinal tap' which involves insertion of a needle into the base of the spinal column in order to extract fluid for diagnostic purposes. The goal is to obtain a fluid sample with minimal trauma on the first attempt. The target space into which the operator is aiming to access this fluid is approx. 3 mm in diameter. First attempt failure rates range from 30-50%. A second try immediately following a first try, even if successful, leads to more trauma to the patient and often a sub-optimal sample (the "bloody tap") due to surrounding tissue/vascular disruption.

Many factors may contribute to first attempt success in this procedure:

1. The clinical condition of the baby including hydration
2. How well pain is controlled (assisting in the reduction of movement)
3. The experience and confidence of the operator conducting the procedure and technique
4. The experience of the assistant positioning the baby. This factor is generally accepted among clinicians as the most important factor contributing to procedure outcome and yet it is highly variable.

The lumbar puncture procedure may be conducted with the baby placed in a side-lying position. The side-lying position is most common, historically, as the patient seems to be more stable. However the alignment of the spine is often disrupted.

The upright sitting position may also be used. There is recent compelling evidence that this position is superior to the side lying position (NeoCLEAR Study 2023)

The sitting position is associated with better outcomes but is often avoided as the holding technique is more complex

The problem which the current innovation seeks to resolve is the high degree of variability in quality, consistency, and reproducibility of a positioning/immobilization of the neonatal patient during the lumbar puncture procedure.

ELIGIBILITY:
Inclusion Criteria:

* Late preterm (34 + weeks) Gestational Age to Term (42+ weeks GA)
* Weight of 2.5 - 5 kg

Exclusion Criteria:

* Any contraindication to having a lumbar punture procedure

Ages: 0 Days to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 68 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
First attempt LP success | Assessed at each procedure
  Primary outcome measure is first attempt LP success (any evidence of CSF which is diagnostically useful by content and volume)

SECONDARY OUTCOMES:
Clear tap | Assessed at each procedure
  A qualitatively unadulterated tap (no blood)
FLACC Score | Assessed at each procedure
  A difference in FLACC score as measure of overall pain/comfort between test and control

CONTACTS AND LOCATIONS:
Overall Officials: Joel B Cox, Medical Doctor, Principal Investigator — Nova Scotia Health Authority

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marshall ASJ, Sadarangani M, Scrivens A, Williams R, Yong J, Bowler U, Linsell L, Chiocchia V, Bell JL, Stokes C, Santhanadass P, Adams E, Juszczak E, Roehr CC; 'The NeoCLEAR Collaborative Group'. Study protocol: NeoCLEAR: Neonatal Champagne Lumbar punctures Every time - An RCT: a multicentre, randomised controlled 2 x 2 factorial trial to investigate techniques to increase lumbar puncture success. BMC Pediatr. 2020 Apr 15;20(1):165. doi: 10.1186/s12887-020-02050-8. PMID 32295554